CLINICAL TRIAL: NCT06223113
Title: Prospective, Registry-based Study to Evaluate Safety and Performance of EyenableTM Intraocular Lens Implantation After Cataract Removal
Brief Title: Evaluation of Safety and Performance of the EyenableTM Intraocular Lens for Cataract Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xi'an Eyedeal Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201-REG
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Cataract
Keywords: Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EyenableTM PA60AS1 IOL implanation (Other): IOL implantation
  Interventions: Device: EyenableTM PA60AS1 IOL

INTERVENTIONS:
Device: EyenableTM PA60AS1 IOL — Subjects will undergo surgery to remove cataract (the cloudy lenses) via phacoemulsification, and implant the Eyedeal® EyenableTM PA60AS1 IOL in the eye capsule.

SUMMARY:
Cataract is characterized by the loss of the normal transparency of the crystalline lens. It is a progressive, chronic disease that affect individuals over the age of 50. It is the leading cause of blindness around the world. The EyenableTM IOL (PA60AS1) is a CE-marked foldable single-piece ultra-violet absorbing posterior chamber intraocular lens (IOL). It is an optical implant to replace the human crystalline lens in the visual correction of aphakia in adult patients after cataract removal. This post-market clinical study will investigate the implantation safety and performance of the EyenableTM PA60AS1 intraocular lens (IOL) up to 6 month after the surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years of age at the time of surgery) of any gender, diagnosed with age related cataracts in one or both eyes.
2. Opacity of crystalline lens due to cataract and reduced vision assessed by patient complaints.
3. Calculated lens power within the available range for the EyenableTM PA60AS1 IOL (+10D to +30.00D)
4. Planned cataract removal by phacoemulsification procedure
5. Clear intraocular media other than cataract, in the study eye
6. Pharmacologically dilated pupil size of at least 6.0mm.
7. 2.0 D or less of preoperative astigmatism in the study eye
8. Willing and able to complete all required postoperative visits
9. Able and willing to comprehend and sign or through a representative, with a witness present, an EC approved Informed Consent Form (ICF).

Exclusion Criteria:

1. Subject who, in the judgment of the clinical investigator, is not suitable for participation in the study for any clinical reason, as documented by the investigator on the patient's Case Report Forms (CRFs).
2. Any type of cataract other than age-related.
3. History of any intraocular, retinal, corneal or refractive surgery in the study eye (including LASIK, PRK, SMILE, etc.), only in the opinion of investigator that it could confound study outcome
4. Ocular conditions which could affect the stability of the IOL (e.g., pseudoexfoliation, zonular dialysis, evident zonular weakness or dehiscence, etc.) in the study eye.
5. Any anterior segment pathology likely to increase the risk of complications from phacoemulsification cataract extraction (e.g., chronic uveitis, iritis, iridocyclitis, aniridia, rubeosis iridis, clinically significant corneal disorders, (Fuchs', or anterior basement membrane dystrophy, etc.) in the study eye.
6. Mature cataract that is likely to prolong phacoemulsification and/or lead to intraoperative complications prior to attempted IOL implantation.
7. Any visually significant intraocular media opacity other than cataract in the study eye.
8. History of any clinically significant retinal pathology or ocular diagnosis (e.g., diabetic retinopathy, ischemic disease, macular degeneration, retinal detachment, amblyopia, optic neuropathy, microphthalmos, aniridia, neuro-ophthalmic disease, fixation problems etc.) in the study eye that could alter or limit final postoperative visual prognosis.
9. History of cystoid macular edema in the study eye.
10. Severe dry eye that, in the opinion of the investigator, would impair the ability to obtain reliable study measurements.
11. Uncontrolled glaucoma and/or optic atrophy in the study eye.
12. Extremely shallow anterior chamber (< 2.0 mm).
13. Irregular astigmatism, corneal degeneration or dystrophy.
14. Uncontrolled systemic disease (e.g., diabetes mellitus, active cancer treatment, mental illness, etc.) in the opinion of the investigator, would put the subject's health at risk and/or prevent the subject from completing all study visits.
15. Systemic medication that, in the opinion of the investigator, may confound the outcome or increase the intraoperative and post-operative risk to the subject (e.g., tamsulosin hydrochloride)
16. Subjects who may reasonably be expected to require any additional ophthalmic surgical intervention at any time during the study (other than YAG capsulotomy).
17. Need for concomitant procedures (e.g., glaucoma surgery, LRI, PRK, LASIK, etc.).
18. Participation in any other drug or device clinical trial within 30 days prior to enrolling this study and/or during study participation.
19. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
SAFETY OUTCOME MEASURE - Adverse event | 6 month after the device implantation.
  The primary safety endpoints include rates of adverse events, loss of CDVA, slit lamp examination, fundus examination, intraocular pressure, device deficiencies.
PERFORMANCE OUTCOME MEASURE - uncorrected distance visual acuity (UCDVA) | 6 month after the device implantation
  Measurement of UCDVA
PERFORMANCE OUTCOME MEASURE - Corrected distance visual acuity (CDVA) | 6 month after the device implantation
  Measurement of CDVA